CLINICAL TRIAL: NCT00064350
Title: A Double Blind Phase II Study of BAY 43-9006 in Patients With Non-Small Cell Lung Cancer Who Have Failed at Least Two Prior Chemotherapy Regimens
Brief Title: Sorafenib in Treating Patients With Refractory Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000315383; E2501 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2012-11-28 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; sorafenib
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Induction then Sorafenib (Experimental): Induction: All patients receive oral sorafenib twice daily on days 1-28. Treatment continues for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease proceed to randomization. Patients with responding disease continue to receive sorafenib for up to 1 year in the absence of disease progression.
  Randomization: Patients with stable disease after the induction treatment were randomized to either the sorafenib arm or the placebo arm. Patients on the sorafenib arm receive sorafenib twice daily for up to 1 year in the absence of disease progression or unacceptable disease.
  Interventions: Drug: Sorafenib
- Induction then Placebo then Sorafenib (Placebo Comparator): Induction: All patients receive oral sorafenib twice daily on days 1-28. Treatment continues for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease proceed to randomization. Patients with responding disease continue to receive sorafenib for up to 1 year in the absence of disease progression.
  Randomization: Patients with stable disease after the induction treatment were randomized to either the sorafenib arm or the placebo arm. Patients on the placebo arm receive oral placebo twice daily for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients on the placebo arm who develop disease progression within 1 year after randomization may cross over to sorafenib arm.
  Interventions: Drug: Sorafenib; Drug: Placebo
- Induction, not randomized (Other): Induction: All patients receive oral sorafenib twice daily on days 1-28. Treatment continues for 2 cycles in the absence of disease progression or unacceptable toxicity.
  Post-induction: Patients with responding disease or disease progression were not randomized in Step 2. Patients with responding disease continue to receive sorafenib for up to 1 year in the absence of disease progression, while patients with disease progression were removed from the study.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Step 1 (induction): Sorafenib was giventwice daily for two cycles to all patients. Patients with progression (PD) discontinued treatment. Those who responded after two cycles continued treatment up to 1 year or until PD. With response after 1 year, patients were given the option to continue treatment until PD. Patients who were stable after the end of induction were then randomized onto Step 2 to either continue sorafenib or receive placebo.
  Step 2 (randomization): Patients with stable disease after induction will be randomized in a double-blinded manner to placebo or sorafenib. If a patient has progressed, the arm will be unblinded. Patients on placebo with PD can then crossover to receive sorafenib; patients with PD on the sorafenib arm will be removed from the study.
  Step 3 (crossover): If patients on placebo progressed within 1 year from randomization, they crossed over to the treatment arm and receive sorafenib for up to 1 year or until PD, unacceptable toxicity, or death.
  Other Names: Nexavar; BAY 43-9006
Drug: Placebo — Patients randomized to the placebo arm in step 2 continued receiving placebo until disease progression or one year from randomization. Placebo was given orally twice a day (BID).
  Arms: Induction then Placebo then Sorafenib

SUMMARY:
RATIONALE: Preclinical studies indicate that sorafenib is a potent inhibitor of Raf kinase in vitro and in vivo, with significant dose-dependent, anti-tumor activity in four different human tumor types including colon, pancreatic, lung, and ovarian. This activity was cytostatic in nature and was maintained if dosing was continued. That is, tumor growth is suspended while the drug is administered but returns to baseline rates when the agent is withdrawn. Therefore, the optimal schedule will be an uninterrupted one. To assess the activity of sorafenib in a timely manner and with a meaningful interpretation, a randomized discontinuation design was adopted in the present trial, conducted in a population who were potentially sensitive to sorafenib.

PURPOSE: This randomized phase II trial is studying sorafenib to see how well it works compared to placebo in treating patients with refractory non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the percent of patients maintaining stable disease or objective response two months after randomization with continued sorafenib treatment, compared to patients switched to placebo.
* To determine progression-free survival, overall survival, and response rate.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to number of prior chemotherapy regimens (2 vs more than 2) and prior epidermal growth factor receptor inhibitor treatment (yes vs no).

* Induction: All patients receive oral sorafenib twice daily on days 1-28. Treatment continues for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease proceed to randomization. Patients with responding disease continue to receive sorafenib for up to 1 year in the absence of disease progression.
* Randomization: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral sorafenib twice daily for up to 1 year in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive oral placebo twice daily for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients who develop disease progression within 1 year after randomization cross over to arm I.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 311 patients will be accrued for this study within approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced non-small cell lung cancer (NSCLC)
* Disease must have progressed after at least 2 prior chemotherapy regimens for NSCLC
* Patients must have measurable or nonmeasurable disease
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 3 times ULN (5 times ULN in patients with liver disease)
* Creatinine less than 1.5 times ULN or calculated creatinine clearance greater than 50 mL/min
* More than 3 weeks since prior chemotherapy, radiotherapy, immunotherapy or other investigational drug use
* Recovered from all prior therapy
* Fertile patients must use effective contraception
* Age >= 18
* ECOG performance status of 0-1

Exclusion Criteria:

* Prior primary or metastatic brain or meningeal tumors unless clinically and radiographically stable and off therapy for at least 2 months
* Active second malignancy
* Clinically evident congestive heart failure, serious cardiac arrhythmias, or symptoms of coronary heart disease
* Prior radiotherapy to the only site of measurable or evaluable disease unless there is evidence of disease progression in that site
* Prior exposure to a ras pathway inhibitor (e.g., farnesyl transferase inhibitor)
* Concurrent medications known to be metabolized by the liver with a narrow therapeutic index, including the following:

  * Ketoconazole
  * Itraconazole
  * Quinidine
  * Digoxin
  * Cyclosporine
  * Ritonavir
  * Grapefruit products
  * Carbamazepine
  * Phenytoin
  * Phenobarbital
* Pregnant or nursing
* Clinically serious active infection
* Medical conditions, substance abuse or psychological/social situation that would preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2004-06-28 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan H. Schiller, MD, Study Chair — Simmons Cancer Center
Locations (141):
- United States (141):
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Morton Hospital & Medical Center, Taunton, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Foote Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Baptist Regional Cancer Center at Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern University Hospital - Zale Lipshy, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was accrued on May 28, 2004.
Groups:
- Induction Then Sorafenib: Induction: All patients receive oral sorafenib twice daily on days 1-28. Treatment continues for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease proceed to randomization.
  Randomization: Patients with stable disease after the induction treatment were randomized to receive either sorafenib or placebo. Patients on the sorafenib arm receive sorafenib twice daily for up to 1 year in the absence of disease progression or unacceptable disease.
  In the study design, only patients on the placebo arm with progressive disease may cross over to receive sorafenib. Due to drug dispensing error, even though some patients actually received straight sorafenib during Step 2 (randomization) treatment, they were thought to be randomized onto the placebo arm upon progression and unblinding (before finding out the fact of the dispensing error). Consequently, these patients were crossed over to Step 3, and there were 10 of them.
- Induction Then Placebo Then Sorafenib: Induction: All patients receive oral sorafenib twice daily on days 1-28. Treatment continues for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease proceed to randomization. Patients with responding disease continue to receive sorafenib for up to 1 year in the absence of disease progression.
  Randomization: Patients with stable disease after the induction treatment were randomized to either the sorafenib arm or the placebo arm. Patients on the sorafenib arm receive sorafenib twice daily for up to 1 year in the absence of disease progression or unacceptable disease. Patients on the placebo arm receive oral placebo twice daily for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients on the placebo arm who develop disease progression within 1 year after randomization may cross over to sorafenib arm.
- Induction, Not Randomized: Induction: All patients receive oral sorafenib twice daily on days 1-28. Treatment continues for 2 cycles in the absence of disease progression or unacceptable toxicity.
  Patients with responding disease continue to receive sorafenib for up to 1 year in the absence of disease progression.
  Randomization: Patients with stable disease after the induction treatment were randomized to either the sorafenib arm or the placebo arm. Patients in this group did not enter Step 2 (randomization part) after the induction phase.
Period: Induction Treatment
Arm/Group | Induction Then Sorafenib | Induction Then Placebo Then Sorafenib | Induction, Not Randomized
Started | 59 | 46 | 237
Treated | 59 | 46 | 228
Eligible and Treated | 59 | 46 | 194
Completed | 51 | 37 | 1
Not Completed | 8 | 9 | 236
Not completed — Disease Progression | 5 | 1 | 110
Not completed — Adverse Event | 0 | 2 | 49
Not completed — Death | 0 | 0 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 21
Not completed — Ineligible or never started treatment | 3 | 6 | 34
Not completed — Other | 0 | 0 | 13
Period: Randomization
Arm/Group | Induction Then Sorafenib | Induction Then Placebo Then Sorafenib | Induction, Not Randomized
Started | 59 | 46 | 0
Treated | 55 | 40 | 0
Eligible and Treated | 50 | 31 | 0
Completed | 33 | 28 | 0
Not Completed | 26 | 18 | 0
Not completed — Adverse Event | 8 | 3 | 0
Not completed — Death | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Ineligible or never started treatment | 9 | 15 | 0
Not completed — Other | 5 | 0 | 0
Period: Cross-Over
Arm/Group | Induction Then Sorafenib | Induction Then Placebo Then Sorafenib | Induction, Not Randomized
Started | 10 | 27 | 0
Treated | 9 | 26 | 0
Eligible and Treated | 7 | 21 | 0
Completed | 4 | 13 | 0
Not Completed | 6 | 14 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Death | 1 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Ineligible or never started treatment | 3 | 6 | 0
Not completed — Other | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Induction, Not Randomized: Induction: All patients receive oral sorafenib twice daily on days 1-28. Treatment continues for 2 cycles in the absence of disease progression or unacceptable toxicity.
  Patients with responding disease continue to receive sorafenib for up to 1 year in the absence of disease progression.
  Randomization: Patients with stable disease after the induction treatment were randomized to either the sorafenib arm or the placebo arm.
  To show baseline characteristics for eligible and treated patients in both the randomization phase (the most important part of this study) and the induction phase, this group contains the following patients:
  * eligible and treated patients who were not randomized (n=194)
  * randomized patients who were not eligible or did not start treatment in the randomization phase (n=24)
  There were 218 patients in this group so the total number of patients is 299 and the entire cohort represents all eligible and treated patients in the induction phase.
- Total: Total of all reporting groups
Arm/Group | Induction Then Sorafenib | Induction Then Placebo Then Sorafenib | Induction, Not Randomized | Total
Number analyzed (Participants) | 50 | 31 | 218 | 299
Age, Continuous [Median (Full Range); unit: years] | 64.5 [42 to 80] | 69 [40 to 86] | 63 [33 to 85] | 64 [33 to 86]
Sex/Gender, Customized [Number; unit: participants]
  Female | 27 | 13 | 90 | 130
  Male | 23 | 18 | 127 | 168
  Unknown | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Maintaining Stable Disease or Objective Response 2 Months After Randomization
Description: Per RECIST Criteria (V1.0):
  Complete Response (CR): disappearance of all target lesions Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions Progressive Disease (PD): >=20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of longest diameter recorded since randomization, or the appearance of new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
Time Frame: Two months after randomization
Measure: Number; unit: participants
Groups:
- Sorafenib: Patients initially received Sorafenib in Step 2 (randomization part)
- Placebo: Patients initially received placebo in Step 2 (randomization part)
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 50 | 31
participants
  Response | 0 | 0
  Stable Disease | 27 | 7
  Progression | 19 | 23
  Unevaluable | 4 | 1
Statistical Analysis 1: Comparison: Sorafenib vs Placebo; Compare the proportion of patients maintaining stable disease or objective response at 2 months after randomization between the two arms; Test type: Superiority or Other; p = 0.005, Fisher Exact

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the duration from randomization to disease progression or death, whichever occurs first. Only randomized patients were included in this analysis.
Time Frame: Assessed every 8 weeks while on treatment. After the end of treatment, assessed every 3 months for 2 years, then every 6 months for 3 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 50 | 31
Months | 3.3 [2.1 to 4.7] | 2.0 [1.8 to 2.3]
Statistical Analysis 1: Comparison: Sorafenib vs Placebo; Compare PFS between the Sorafenib arm and the placebo arm; Test type: Superiority or Other; p = 0.014, Log Rank

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration from randomization to death or last known alive. Only randomized patients were included in this analysis.
Time Frame: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 50 | 31
Months | 13.7 [7.9 to 17.8] | 9.0 [6.7 to 11.7]
Statistical Analysis 1: Comparison: Sorafenib vs Placebo; Compare OS between the Sorafenib arm and the placebo arm; Test type: Superiority or Other; p = 0.12, Log Rank

4. Secondary Outcome: Best Overall Response
Description: The best overall response is the best response (per RECIST 1.0) recorded from randomization until disease progression/recurrence, taking as reference for progressive disease the smallest measurements recorded since randomization.
Time Frame: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 50 | 31
Participants
  Complete Response | 0 | 0
  Partial Response | 1 | 1
  Stable Disease | 28 | 6
  Progression | 20 | 24
  Unevaluable | 1 | 0

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 28 days after the end of treatment
Groups:
- Induction: Sorafenib: All patients who received induction treatment (333 patients), regardless of eligibility status, were included in the toxicity analysis.
- Randomization (Step 2): Sorafenib: After induction treatment, 59 patients were randomized to the sorafenib arm. Among these, 55 received treatment. However, due to drug dispensing error, 10 of them received mixed treatment with sorafenib and placebo and were categorized into "Randomization (Step 2): Mixed" group when reporting toxicities. As a result, 45 treated patients were included in the "randomization (step 2): sorafenib" group.
- Randomization (Step 2): Placebo: After induction treatment, 46 patients were randomized to the placebo arm. Among these, 40 received treatment. However, due to drug dispensing error, 2 of them received mixed treatment with sorafenib and placebo and were categorized into "Randomization (Step 2): Mixed" group when reporting toxicities. As a result, 38 treated patients were included in the "randomization (step 2): placebo" group.
- Randomization (Step 2): Mixed: After induction treatment, patients with stable disease were randomized to receive either sorafenib or placebo. Due to drug dispensing error, 10 patients from the sorafenib arm and 2 patients from the placebo arm (12 pts in total) received mixed treatment with sorafenib and placebo and were categorized into "Randomization (Step 2): Mixed" group when reporting toxicities.
- Crossover: Sorafenib: Patients on the placebo arm who develop progressive disease may cross over to receive sorafenib, and 27 patients from the placebo arm received sorafenib in Step 3 (crossover). Due to drug dispensing error, even though some patients actually received straight sorafenib during Step 2 (randomization) treatment, they were thought to be randomized onto the placebo arm upon progression and unblinding (before finding out the fact of the dispensing error). Consequently, these patients were crossed over to Step 3, and there were 10 of them. In total, 37 patients registered to step 3 (crossover). Of these, 35 patients received treatment and were included in the toxicity analysis for the crossover (step 3) part.
Arm/Group | Induction: Sorafenib | Randomization (Step 2): Sorafenib | Randomization (Step 2): Placebo | Randomization (Step 2): Mixed | Crossover: Sorafenib
Serious Adverse Events (participants affected / at risk) | 133/333 | 16/45 | 7/38 | 2/12 | 15/35
Other Adverse Events (participants affected / at risk) | 307/333 | 42/45 | 34/38 | 11/12 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction: Sorafenib (N=333) | Randomization (Step 2): Sorafenib (N=45) | Randomization (Step 2): Placebo (N=38) | Randomization (Step 2): Mixed (N=12) | Crossover: Sorafenib (N=35)
ALT increased (Investigations) | 1 | 0 | 0 | 0 | 0
AST increased (Investigations) | 2 | 0 | 0 | 0 | 0
Abdomen, pain (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 2
Alkaline phosphatase increased (Investigations) | 2 | 1 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 2 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 10 | 0 | 1 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 0 | 1
Bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Bone, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 4 | 1 | 0 | 0 | 0
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Chest/thoracic pain NOS (General disorders) | 3 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Death - disease progression NOS (General disorders) | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5 | 2 | 0 | 0 | 2
Distention/bloating, abdominal (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 1 | 1 | 1 | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 35 | 3 | 2 | 1 | 6
GGT (Investigations) | 0 | 1 | 0 | 0 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 32 | 2 | 0 | 0 | 0
Head/headache (Nervous system disorders) | 5 | 0 | 0 | 0 | 0
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 10 | 1 | 1 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
INR (Investigations) | 6 | 3 | 1 | 0 | 0
Infection - other (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Infection with Grade 0-2 neutropenia, lung (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection with Grade 3-4 neutropenia, lung (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection with unknown ANC, lung (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Lymphopenia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Muco/stomatitis (symptom), oral cavity (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 1 | 0 | 0 | 2
Neurologic - other (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy - motor (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Neuropathy - sensory (Nervous system disorders) | 4 | 0 | 0 | 0 | 1
Neutropenia (Investigations) | 2 | 0 | 0 | 0 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Ocular - other (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Oral gums, pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Prolonged QTc interval (Investigations) | 1 | 0 | 0 | 0 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 21 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Respiratory tract hemorrhage NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Speech impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Stomach, pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Investigations) | 2 | 0 | 0 | 0 | 0
Thrombosis/embolism (Vascular access-related) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thrombosis/thrombus/embolism (Injury, poisoning and procedural complications) | 8 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction: Sorafenib (N=333) | Randomization (Step 2): Sorafenib (N=45) | Randomization (Step 2): Placebo (N=38) | Randomization (Step 2): Mixed (N=12) | Crossover: Sorafenib (N=35)
Anemia (Blood and lymphatic system disorders) | 96 | 16 | 15 | 3 | 17
Leukopenia (Investigations) | 35 | 5 | 1 | 1 | 6
Thrombocytopenia (Investigations) | 36 | 4 | 5 | 0 | 6
Hypertension (Vascular disorders) | 28 | 6 | 1 | 0 | 1
Fatigue (General disorders) | 156 | 24 | 16 | 7 | 20
Weight loss (Investigations) | 37 | 5 | 5 | 2 | 7
INR increased (Investigations) | 20 | 4 | 2 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 32 | 8 | 2 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 11 | 1 | 1 | 5
Pruritus/itching (Skin and subcutaneous tissue disorders) | 56 | 6 | 1 | 1 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 115 | 18 | 9 | 7 | 10
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 48 | 10 | 2 | 3 | 5
Anorexia (Metabolism and nutrition disorders) | 104 | 16 | 6 | 2 | 9
Constipation (Gastrointestinal disorders) | 30 | 8 | 0 | 1 | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 87 | 15 | 5 | 9 | 19
Dyspepsia (Gastrointestinal disorders) | 30 | 4 | 2 | 1 | 3
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 28 | 2 | 1 | 0 | 1
Muco/stomatitis (symptom), oral cavity (Gastrointestinal disorders) | 39 | 3 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 65 | 12 | 6 | 2 | 13
Vomiting (Gastrointestinal disorders) | 33 | 6 | 3 | 0 | 4
Alkaline phosphatase increased (Investigations) | 73 | 10 | 6 | 2 | 7
ALT increased (Investigations) | 26 | 7 | 6 | 1 | 5
AST increased (Investigations) | 50 | 12 | 5 | 2 | 10
Neuropathy - sensory (Nervous system disorders) | 30 | 5 | 1 | 2 | 3
Head/headache (Nervous system disorders) | 24 | 6 | 1 | 0 | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 20 | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 4 | 4 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 | 6 | 4 | 0 | 3
Lymphopenia (Investigations) | 5 | 0 | 0 | 0 | 2
Fever w/o neutropenia (General disorders) | 7 | 0 | 1 | 0 | 2
Rigors/chills (General disorders) | 3 | 0 | 0 | 0 | 4
Flushing (Vascular disorders) | 12 | 0 | 2 | 0 | 3
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 8 | 1 | 0 | 1 | 3
Flatulence (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 4
Taste disturbance (Gastrointestinal disorders) | 13 | 3 | 1 | 2 | 2
Bilirubin increased (Investigations) | 14 | 1 | 1 | 1 | 2
Creatinine increased (Investigations) | 7 | 1 | 4 | 0 | 2
Abdomen, pain (Gastrointestinal disorders) | 10 | 2 | 4 | 0 | 3
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 16 | 1 | 0 | 1 | 2
Back, pain (Musculoskeletal and connective tissue disorders) | 11 | 4 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 1 | 1 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 0 | 1 | 0
Wound - non-infectious (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0
Incontinence, anal (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Infection Grade 0-2 neutropenia, upper airway (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Edema head and neck (General disorders) | 8 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 10 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 5 | 1 | 0 | 1 | 1
Neuropathy - motor (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Oral cavity, pain (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 0
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No